CLINICAL TRIAL: NCT06019546
Title: Perfusion Quality Odds
Acronym: PEQUOD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Marco Ranucci, Director of the Cardiovascular Anesthesia and Intensive Care Department, IRCCS Policlinico S. Donato
Other Study IDs: PEQUOD
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cardiac Disease; Extracorporeal Circulation; Complications; Perfusion; Complications; Acute Kidney Injury
Keywords: acute kidney injury; cardiopulmonary bypass; cardiac surgery; risk score
MeSH Terms: conditions — Heart Diseases; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PEQUOD: Patients undergoing cardiac surgery with cardiopulmonary bypass whose parameters of interest will be registered during cardiopulmonary bypass by the Livanova BE-CAPTA monitor.
  Interventions: Other: PEQUOD

INTERVENTIONS:
Other: PEQUOD — During cardiopulmonary bypass registration of the parameters of interest by the Livanova BE-CAPTA monitor. After surgery, registration of creatinine values up to 48 postoperative hours.

SUMMARY:
Cardiac surgery-associated acute kidney injury (CSA-AKI) is a frequent complication after cardiac operations with cardiopulmonary bypass (CPB) use. Its frequency varies depending on the severity grade. There are different "static" predictive scores for the CSA-AKI based on the patient and surgery-associated parameters.

Recently, in our Institution was developed a predictive algorithm for CSA-AKI that starts with a static model and then integrated with 7 CPB-associated parameters: HCT, DO2, time of exposure to a critical DO2, systemic pressure, CPB duration time, lactate value, transfusion of red blood cells (RBC), that together build a dynamic perfusion risk (DPR) associated to the CPB. Combining the static and dynamic models produces the Multifactorial Dynamic Perfusion Index (MDPI).

The present study validates MDPI in a new prospective series of patients undergoing cardiac surgery with CPB.

DETAILED DESCRIPTION:
Cardiac surgery-associated acute kidney injury (CSA-AKI) is a frequent complication after cardiac operations with cardiopulmonary bypass (CPB) use. Its frequency varies depending on the severity grade which for the present study follows the AKIN criteria.

There are different predictive scores for the CSA-AKI based on the patient and surgery-associated parameters. These models could be defined as "static".

It's known that a number of CPB-associated parameters could influence CSA-AKI, as well. These include hematocrit (HCT), oxygen delivery (DO2), time of exposure to a critical DO2, and perfusion pressure. These parameters, taken separately, are associated with CSA-AKI development.

Recently, our Institution has developed a predictive algorithm for CSA-AKI that starts with a static model and then integrated with 7 CPB-associated parameters: HCT, DO2, time of exposure to a critical DO2, systemic pressure, CPB duration time, lactate value, transfusion of red blood cells (RBC), that together build a dynamic perfusion risk (DPR) associated to the CPB. Combining the static and dynamic models produces the Multifactorial Dynamic Perfusion Index (MDPI).

MDPI has higher discrimination power when compared to the static scores, in the original series and in the internal validation with the Bootstrap technique.

The present study validates MDPI in a new prospective series of patients undergoing cardiac surgery with CPB. An enrollment of 400 patients is anticipated with a stopping rule for efficacy at interim analysis (for primary endpoint) at 50% enrollment (200 patients) if the c-statistics for any stage of CSA-AKI reaches at least 0.75. Futility is defined as an AUC of 0.6 or lower.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cardiac surgery with cardiopulmonary bypass
* age of 18 years and higher
* willingness to participate and sign the informed consent

Exclusion Criteria:

- patients requiring preoperative dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in our Institution for a scheduled cardiac surgery with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with postoperative acute kidney injury | First 48 postoperative hours
  Occurence of any stage acute kidney injury as defined by the AKIN criteria

SECONDARY OUTCOMES:
Number of patients with postoperative respiratory insufficiency | First 48 postoperative hours
  P/F ratio > 200 with radiographic evidence of pulmonary distress, if compared to the baseline by an independent radiologist
Number of patients with postoperative low cardiac output | First 48 postoperative hours
  Use of inotrope drugs for more than 48 hours and/or mechanical support
Number of patients experiencing postoperative major morbidity | First 48 postoperative hours
  As defined by STS criteria as one or more of the following items: AKI stage 2, stroke, mechanical ventilation duration > 48 hours, sepsis, surgical re-exploration
Number of patients who needed prolonged ICU stay | First 4 postoperative days
  ICU stay duration > 4 days
Number of deceased patients | 30 days after surgery
  Dead or alive status

CONTACTS AND LOCATIONS:
Overall Officials: Marco Ranucci, MD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, MI, Italy

IPD SHARING:
Plan to Share IPD: No
The original dataset supporting the findings of this study will be deposited in the public repository Zenodo after the publication of the work and accessible upon a reasonable request. The requests should be addressed to the Principal Investigator of the study.

REFERENCES:
- [Background] Ranucci M, Aloisio T, Cazzaniga A, Di Dedda U, Gallazzi C, Pistuddi V. Validation of renal-risk models for the prediction of non-renal replacement therapy cardiac surgery-associated acute kidney injury. Int J Cardiol. 2018 Dec 1;272:49-53. doi: 10.1016/j.ijcard.2018.07.114. Epub 2018 Jul 24. PMID 30078648
- [Background] Thakar CV, Arrigain S, Worley S, Yared JP, Paganini EP. A clinical score to predict acute renal failure after cardiac surgery. J Am Soc Nephrol. 2005 Jan;16(1):162-8. doi: 10.1681/ASN.2004040331. Epub 2004 Nov 24. PMID 15563569
- [Background] Mehta RH, Grab JD, O'Brien SM, Bridges CR, Gammie JS, Haan CK, Ferguson TB, Peterson ED; Society of Thoracic Surgeons National Cardiac Surgery Database Investigators. Bedside tool for predicting the risk of postoperative dialysis in patients undergoing cardiac surgery. Circulation. 2006 Nov 21;114(21):2208-16; quiz 2208. doi: 10.1161/CIRCULATIONAHA.106.635573. Epub 2006 Nov 6. PMID 17088458
- [Background] Wijeysundera DN, Karkouti K, Dupuis JY, Rao V, Chan CT, Granton JT, Beattie WS. Derivation and validation of a simplified predictive index for renal replacement therapy after cardiac surgery. JAMA. 2007 Apr 25;297(16):1801-9. doi: 10.1001/jama.297.16.1801. PMID 17456822
- [Background] Swaminathan M, Phillips-Bute BG, Conlon PJ, Smith PK, Newman MF, Stafford-Smith M. The association of lowest hematocrit during cardiopulmonary bypass with acute renal injury after coronary artery bypass surgery. Ann Thorac Surg. 2003 Sep;76(3):784-91; discussion 792. doi: 10.1016/s0003-4975(03)00558-7. PMID 12963200
- [Background] Habib RH, Zacharias A, Schwann TA, Riordan CJ, Durham SJ, Shah A. Adverse effects of low hematocrit during cardiopulmonary bypass in the adult: should current practice be changed? J Thorac Cardiovasc Surg. 2003 Jun;125(6):1438-50. doi: 10.1016/s0022-5223(02)73291-1. PMID 12830066
- [Background] Ranucci M, Romitti F, Isgro G, Cotza M, Brozzi S, Boncilli A, Ditta A. Oxygen delivery during cardiopulmonary bypass and acute renal failure after coronary operations. Ann Thorac Surg. 2005 Dec;80(6):2213-20. doi: 10.1016/j.athoracsur.2005.05.069. PMID 16305874
- [Background] Ranucci M, Johnson I, Willcox T, Baker RA, Boer C, Baumann A, Justison GA, de Somer F, Exton P, Agarwal S, Parke R, Newland RF, Haumann RG, Buchwald D, Weitzel N, Venkateswaran R, Ambrogi F, Pistuddi V. Goal-directed perfusion to reduce acute kidney injury: A randomized trial. J Thorac Cardiovasc Surg. 2018 Nov;156(5):1918-1927.e2. doi: 10.1016/j.jtcvs.2018.04.045. Epub 2018 Apr 18. PMID 29778331
- [Background] Rasmussen SR, Kandler K, Nielsen RV, Cornelius Jakobsen P, Knudsen NN, Ranucci M, Christian Nilsson J, Ravn HB. Duration of critically low oxygen delivery is associated with acute kidney injury after cardiac surgery. Acta Anaesthesiol Scand. 2019 Nov;63(10):1290-1297. doi: 10.1111/aas.13457. Epub 2019 Sep 10. PMID 31436307
- [Background] de la Hoz MA, Rangasamy V, Bastos AB, Xu X, Novack V, Saugel B, Subramaniam B. Intraoperative Hypotension and Acute Kidney Injury, Stroke, and Mortality during and outside Cardiopulmonary Bypass: A Retrospective Observational Cohort Study. Anesthesiology. 2022 Jun 1;136(6):927-939. doi: 10.1097/ALN.0000000000004175. PMID 35188970
- [Background] Ranucci M, Di Dedda U, Cotza M, Zamalloa Moreano K. The multifactorial dynamic perfusion index: A predictive tool of cardiac surgery associated acute kidney injury. Perfusion. 2024 Jan;39(1):201-209. doi: 10.1177/02676591221137033. Epub 2022 Oct 28. PMID 36305847